CLINICAL TRIAL: NCT04857411
Title: Improving Diabetes Programs for Blacks in Wisconsin: Peers as Coaches in Medicine Use
Brief Title: Peers LEAD Plus Healthy Living With Diabetes (HLWD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-1061; A561000 (Other: UW Madison); PHARM/PHARMACY (Other: UW Madison); Protocol Version 2/24/2021 (Other: UW Madison); Baldwin Grant (Other: UW Office of the Provost)
Record Dates: First submitted 2021-04-22; First posted 2021-04-23 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Medication adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant 'Buddies' (Experimental): Participants will have an 8-week program initiation phase followed by a maintenance phase through 6-months, supported by Ambassadors.
  Interventions: Behavioral: Peers LEAD plus HLWD

INTERVENTIONS:
Behavioral: Peers LEAD plus HLWD — Combined Peers LEAD and Healthy Living with Diabetes is a culturally-appropriate program to increase medication adherence

SUMMARY:
The specific goal of this project is to decrease diabetes-related morbidity among African Americans (AAs) in Milwaukee through the integration of Peers LEAD, a culturally-appropriate program to increase medication adherence into Healthy Living with Diabetes (HLWD), an existing diabetes self-management program.

DETAILED DESCRIPTION:
This project represents the next phase of prior work at the University of Wisconsin School of Pharmacy to create and implement community-based programs for AAs with diabetes that focus on improving medication use and glycemic control. The overall objective is to integrate Peers LEAD into HLWD using a community-engaged approach and an evaluation to document outcomes. This project will produce a culturally-tailored curriculum that can be used broadly across social service and community organizations, faith-based organizations, and federally-qualified health centers committed to improving AAs diabetes self-management. This project will be achieved through the following objectives:

* Objective 1: To gather and incorporate key stakeholders input in the current and future adoption of Peers LEAD+HLWD into community organizations, health system and/or practices. Objective 1 is not a clinical trial.
* Objective 2: To implement and measure the outcomes of Peers LEAD+HLWD to improve medication adherence and hemoglobin A1c. Objective 2 represents the clinical trial aim of this study to be registered in this record.

HLWD is a successful community-based program that offers tools and resources to enhance understanding of what it means to have diabetes, including helping participants to build the confidence to manage diabetes and maintain an active and fulfilling life. HLWD is endorsed by the American Diabetes Association and the Centers for Disease Prevention and Control and proven to reduce emergency department visits by 53%, improve A1c levels, enhance regular treatment and diabetes education, create a community-clinical link in care, provide social benefits for participants, improve self-rated health and communication with physicians, and improve health status, health behavior, and self-efficacy. The investigators chose HLWD as the diabetes self-management education (DSME) program to adapt because it is an effective and widely-disseminated evidence-based DSME program. HLWD has enrolled over 5,000 participants in more than 400 workshops across 52 Wisconsin counties. However, between 2013 and 2016, only 120 AAs (3.1%) participated compared to 1,656 non-Hispanic Whites. In 3 years, only 46% of AAs reported that they took their diabetes pills (HLWD's measure of medication adherence) after the workshop, compared to 55% of non-Hispanic Whites. Despite HLWD's positive outcomes and wide reach, there is limited inclusion of AAs. HLWD does not offer culturally-tailored content for AAs, and lacks one-on-one peer support from an AA who successfully manages diabetes, an important factor influential in improving diabetes outcomes among AAs. There is also insufficient attention to medication adherence. Adding Peers LEAD to HLWD will improve the reach, effectiveness, and impact of diabetes self-management programs among AAs.

Peers LEAD is a culturally-tailored program designed to provide AAs with diabetes and medication beliefs information, behavioral skill-development, and one-on-one peer support to increase medication adherence. Group sessions include discussions of personal discrimination experiences that resulted in provider mistrust, making the most of clinic/pharmacy visits, necessity and concerns about medicines, and enhancing patient-provider communication. Ambassadors are paired with Buddies, and Ambassadors help deliver Peers LEAD content via face-to-face interaction with their Buddies during group sessions and phone follow-ups. Ambassadors address misperceptions of medicines and diabetes, share their experiences managing diabetes and medicines, and discuss building relationships with providers. As well, they are able to provide one-on-one social support.

Peers LEAD+HLWD allows for sufficient attention to medication adherence in a DSME program. For example, HLWD includes only one 20-minute activity on medication use in a 2½ hour session during Week 5. This activity only covers purpose of medicines, medication effects, and remembering to take medicines, but does not address known specific barriers to AAs adherence. In this study, HLWD will be adapted for AAs by adding components of Peers LEAD to overcome key barriers to AAs medication adherence. Core components of Peers LEAD to be incorporated are two group sessions on beliefs about medicines and diabetes, discrimination/mistrust, and provider communication, as well as peer-based phone support from Ambassadors.

The investigators hypothesize that, by implementing Peers LEAD+HLWD, there will be increased reach, engagement, and impact for AAs because psychosocial/sociocultural factors and barriers identified in their work to influence AAs medication adherence (i.e., culturally embedded health beliefs and provider mistrust) will be addressed.

Objective 2 is a pre-post single group design to conduct Peers LEAD+HLWD in Milwaukee. There will be two groups of participants: (1) Ambassadors (who are not consented into the intervention, but help facilitate it) - AAs who have diabetes and are adherent with their medicines and (2) Buddies (consented into the intervention) - who are AAs who have diabetes but are nonadherent with their medicines.

Training of Ambassadors: To prepare to implement Peers LEAD+HLWD, Ambassadors will attend a 6-hour orientation and training meetings, co-facilitated by Wisconsin Network for Research Support (WINRS). This meeting will be an orientation and will prepare the Ambassadors to implement specific elements of Peers LEAD+HLWD, such as the phone calls. WINRS will consult with the research team on all meetings. For >8 years, WINRS staff have been deeply involved in stakeholder engagement, as well as trained, planned and facilitated >250 lay advisory board meetings.

Ambassadors are involved in two group sessions focusing on beliefs about medicines and diabetes, discrimination/mistrust, and communication with providers, and peer-based phone support with buddies to occur weekly for the first 2 weeks, then for 5 weeks after the completion of the 8-week program. Building on the previously piloted version of Peers LEAD, Peers LEAD + HLWD has added phone-based peer support from Ambassadors comprised of bi-weekly calls to monitor progress toward goals (Month 4) and finally monthly calls to support goal adherence (Months 5-6), representing the Maintenance Phase.

ELIGIBILITY:
Shared Inclusion Criteria for Ambassadors and Buddies:

* Self-identify as AA
* Can speak/read English
* Self-report being prescribed one oral or injectable diabetes medication
* Access to/can use a cellular phone, tablet or computer to join a web-based meeting by video camera during the study period
* Diagnosed with diabetes for ≥1 year (obtained by self-report or verified by electronic medical record)
* Will reside in the geographical area throughout the study period

Inclusion Criteria Specific to Buddies:

* Self-reported nonadherence on the Adherence to Reﬁlls and Medications Scale for Diabetes (ARMS-D) scale
* Most recent A1c is ≥8% based on information collected at point of care A1c testing

Inclusion Criteria Specific to Ambassadors:

* Self-reported adherence on the Adherence to Reﬁlls and Medications Scale for Diabetes (ARMS-D) scale
* Most recent A1c is <8% based on point of care A1c test
* Willing to provide support to a Buddy and track phone conversations
* Willing to attend all training sessions and meetings related to being an Ambassador

Shared Exclusion Criteria for Ambassadors and Buddies:

* Diagnosed psychiatric disorder
* Older than 65-years old with a history of severe hypoglycemia requiring medical assistance or glucagon administration

Exclusion Criteria Specific to Buddies:

* Currently participating in another diabetes lifestyle self-management or medication adherence program

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Mean Hemoglobin A1c | baseline
  Participant buddies will have a hemoglobin A1c greater than 8 percent at baseline. will be measured using the A1cNow+ system, the National Glycohemoglobin Standardization Program Certified, CLIA-waived, system that provides results using a finger stick test.
Mean Hemoglobin A1c | 3 months
  Participant buddies will have a hemoglobin A1c greater than 8 percent at baseline. will be measured using the A1cNow+ system, the National Glycohemoglobin Standardization Program Certified, CLIA-waived, system that provides results using a finger stick test.
Mean Hemoglobin A1c | 6 months
  Participant buddies will have a hemoglobin A1c greater than 8 percent at baseline. will be measured using the A1cNow+ system, the National Glycohemoglobin Standardization Program Certified, CLIA-waived, system that provides results using a finger stick test.
Mean Systolic Blood Pressure | baseline
  Blood pressure readings collected via the Omron Healthcare Inc. 7 Series Upper Arm Blood Pressure Monitor.
Mean Systolic Blood Pressure | 3 months
  Blood pressure readings collected via the Omron Healthcare Inc. 7 Series Upper Arm Blood Pressure Monitor.
Mean Systolic Blood Pressure | 6 months
  Blood pressure readings collected via the Omron Healthcare Inc. 7 Series Upper Arm Blood Pressure Monitor.
Change in Diastolic Blood Pressure | baseline, 3 months, 6 months
  Blood pressure readings collected via the Omron Healthcare Inc. 7 Series Upper Arm Blood Pressure Monitor.

SECONDARY OUTCOMES:
Adherence to Reﬁlls and Medications Scale for Diabetes (ARMS-D) Score | baseline, 3 months, 6 months
  ARMS-D is a measure of medication adherence. It is an 11-item survey with a total possible range of scores 11-44. Lower scores indicate better medication adherence.
Self-Efficacy for Adherence to Medication Use Scale (SEAMS) | baseline, 3 months, 6 months
  SEAMS is a 16-item questionnaire that assesses peoples' confidence in taking their medications correctly, which can be used to determine medication self-efficacy in a person with diabetes. Current evidence exists demonstrating the reliability and validity of the SEAMS instrument. Respondents are asked to indicate, under a number of different circumstances, their level of confidence about taking medications correctly. Each item is evaluated using a 3-point Likert-type scale (1 = not confident, 2 = somewhat confident, and 3 = very confident). The sum of SEAMS ranges from 13 to 39. Higher scores reflect that respondents have more confidence in being adherent to their medication use.
Patient's Perceived Involvement in Care Scale (PICS) | baseline, 3 months, 6 months
  PICS is a brief, psychometrically-sound, self-report questionnaire about primary care patients' attitudes regarding their illnesses and the management of them. This instrument is designed to examine three relatively distinct factors: (1) doctor facilitation of patient involvement, (2) level of information exchange, and (3) patient participation in decision making.
  This instrument evaluates doctor-patient interactions across three relatively distinct factors, including doctor facilitation of patient involvement (5 items), level of information exchange (4 items), and patient participation in decision making (4 items). In total, respondents answer 13 dichotomous items (0 point is given for "no" and 1 point for "yes.") Items scores are summed to generate a total score ranging from 0-13, and higher scores suggest a greater degree of shared decision making for disease self-management.
Diabetes Distress Scale (DDS) 2 | baseline, 3 months, 6 months
  The DDS-2 is a 2-item screener version of the reliable and valid 17-item DDS questionnaire, which is constructed for people with type 2 diabetes. The DDS-2 is a simple method to evaluate peoples' feelings about being overwhelmed by the demands of living with diabetes and about the extent that people believe that they are failing with their diabetes routine. Each item is evaluated using a 6-point scale (1 and 2 = not a problem, 3 and 4 = moderate problem, and 5 and 6 = serious problem) for a range of possible scores between 2 and 12. People who rate these two items higher are reporting a greater the degree to which diabetes-related distress is bothering them in their lives.
Patient Health Questionnaire (PHQ-4) | baseline, 3 months, 6 months
  PHQ-4 is an 4-item instrument that is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies, and also serves as a useful measure for the purpose of population-based studies. A score of 10 or greater is considered major depression, 20 or more is severe major depression.
Diabetes Empowerment Scale - Short Form (DES-SF) | baseline, 3 months, 6 months
  The DES-SF is an 8-item short form of the original 37-item Diabetes Empowerment Scale. The DES-SF allows for a brief overall assessment of diabetes-related psychosocial self-efficacy. Investigations have provided preliminary evidence that the DES-SF is a valid and reliable measure of overall diabetes-related psychosocial self-efficacy.
  An item checked "strongly agree" receives 5 points; "agree" - 4 points; "neutral" - 3 points; "disagree" - 2 points; and "strongly disagree" receives 1 point. The possible range of scores is 8-40, with higher scores indicating higher diabetes-related psychosocial self-efficacy.
Brief Illness Perception Questionnaire (Brief IPQ) | baseline, 3 months, 6 months
  The Brief IPQ is a 9-item questionnaire designed to rapidly assess cognitive and emotional representations of illness. The Brief IPQ uses a single-item scale approach to assess perception on a 0-10 continuous linear response scale. Overall, the Brief IPQ is a psychometrically sound instrument that provides a rapid assessment of illness perceptions, and can be particularly helpful in ill populations, large-scale studies, and in repeated measures research designs.
  To compute the score, reverse score items 3, 4, and 7 and add these to items 1, 2, 5, 6, and 8 for a range of scores from 0-80. A higher score reflects a more threatening view of the illness. Item 9 is qualitative and not scored with the other items. It asks respondents to list in rank-order the three most important factors they believe caused their illness.
Beliefs about Medicines Questionnaire (BMQ) | baseline, 3 months, 6 months
  The BMQ is a tool for evaluating people's beliefs about the necessity of medications and concerns about using those medications. It has been validated for use in patients with chronic illnesses and has been shown to predict adherence to treatment among people with type 2 diabetes.
  The BMQ has 10-items and consists of two 5-item subscales: necessity beliefs and concern beliefs. Each item is measured on 5-point Likert-type scales with 'strongly disagree (score = 1)' to 'strongly agree (score = 5)' response options. The scores summed for each subscale range from 5-25, with a higher score meaning stronger necessity or concern beliefs about the medication prescribed for personal use.
Newest Vital Sign (NVS) | baseline, 3 months, 6 months
  The NVS is a 6-item assessment of respondent's health literacy in the following areas: literacy, comprehension, application/function, evaluation, and numeracy skills. Each question is scored "0" for incorrect and "1" for correct yielding a total score ranging from 0 to 6, with higher scores indicating better health literacy. Scores of less than 2 represents high likelihood (50% or more) of limited (inadequate) literacy, 2 to 3 indicates possibility of limited (marginal) literacy, and more than 3 suggests adequate literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Olayinka Shiyanbola, PhD, B.Pharm, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Community Locations, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shiyanbola OO, Maurer M, Schwerer L, Sarkarati N, Wen MJ, Salihu EY, Nordin J, Xiong P, Egbujor UM, Williams SD. A Culturally Tailored Diabetes Self-Management Intervention Incorporating Race-Congruent Peer Support to Address Beliefs, Medication Adherence and Diabetes Control in African Americans: A Pilot Feasibility Study. Patient Prefer Adherence. 2022 Oct 25;16:2893-2912. doi: 10.2147/PPA.S384974. eCollection 2022. PMID 36317056
- See also: UniteWI — https://www.weareunitewi.org/